CLINICAL TRIAL: NCT05035056
Title: Effect of Intensive Medical Treatment on Quantified Coronary Artery Plaque Components With Serial Coronary CTA in Women With NonObstructive CAD
Brief Title: WARRIOR Ancillary Study for CCTA Analysis
Status: Recruiting | Type: Observational
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Damini Dey, Professor and Scientist, Director of Quantitative Image Analysis, Biomedical Imagng Research Institute, Cedars-Sinai Medical Center
Other Study IDs: STUDY00000896; 1R01HL151266 (NIH)
Record Dates: First submitted 2021-08-20; First posted 2021-09-05 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Coronary Artery Disease; Non-Obstructive Coronary Atherosclerosis; Ischemia
MeSH Terms: conditions — Coronary Artery Disease; Ischemia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CT Coronary Angiogram with quantitative characterization of plaque: Participants (102) from Intensive Medical Therapy [IMT] and 102 from the Usual Care [UC] group in the WARRIOR trial) will undergo CTA at the Year 3 follow-up visit (can be as early as 2 years from randomization) at their respective enrollment study sites. Quantitative characterization of plaque analysis will be conducted at Cedars-Sinai Medical Center using Autoplaque plaque analysis software.

SUMMARY:
In this study, quantitative characterization of plaque using coronary computed tomographic angiography (CTA) will be used to determine if women who were treated with intensive medical therapy have a greater reduction in the amount and type of cholesterol plaque compared to women receiving usual care and if this results in beneficial changes in clinical symptoms. The study will provide an understanding of how intensive medical therapy works in providing clinical benefit in women with nonobstructive plaque.

DETAILED DESCRIPTION:
This is an ancillary substudy of the WARRIOR Trial (NCT03417388), a multi-site, PROBE design, that will evaluate an intensive statin/ACE-I (or ARB)/aspirin treatment strategy (IMT) vs. primary prevention risk factor therapy treatment strategy (UC) in 4,422 symptomatic (chronic angina or equivalent) women with non-obstructive CAD (<50% diameter narrowing).

In this ancillary substudy, 204 patients will be recruited from the WARRIOR trial with 102 patients from each of the treatment groups (IMT vs UC). From this cohort, 102 patients per treatment group, most compliant with WARRIOR protocol will undergo a CTA from any time from 2 years post-randomization up to the end of the main WARRIOR study; with changes in plaque and PCAT characteristics quantified.

The main aims are as follows:

1. To compare changes in coronary plaque characteristics and their hemodynamic significance using CTA in WARRIOR women treated with IMT vs UC;
2. To compare changes in plaque inflammation-related characteristics in PCAT in WARRIOR women treated with IMT with statin in combination with angiotensin converting enzyme inhibitor (ACEI) and/or angiotensin receptor blocker (ARB) medications vs UC;
3. To relate plaque burden and plaque composition, CT flow reserve, and PCAT density changes to angina score (Seattle Angina Questionnaire [SAQ]) changes in IMT and UC-randomized WARRIOR women.

Data to be analyzed include CT angiography scans at baseline and Year 3 follow-up and corresponding study data and laboratory tests (e.g. hsCRP); plus, selected data from the main WARRIOR study that are relevant to the present ancillary study.

UPDATE; In this ancillary study, 204 patients will be recruited from the WARRIOR Trial with 102 patients from each of the treatment groups (IMT vs UC). From this cohort, 102 patients per treatment group, most compliant with WARRIOR protocol will undergo a CTA as early as 2 years after their randomization to the WARRIOR trial up to study completion; with changes in plaque and CAT characteristics quantified.

ELIGIBILITY:
Inclusion Criteria:

* In addition to the inclusion criteria of the WARRIOR trial, only women who meet the following criteria will undergo final CTA at the same sites where they are screened and enrolled.
* Initial CTA with excellent or good image quality-defined as images where we are able to clearly identify the atherosclerotic plaque. Based on our preliminary assessment, we expect 90% of studies to be included.
* Measurable plaque with total plaque volume >0mm3; women without significant plaque will not receive additional radiation, and we can detect measurable changes in plaque burden and plaque composition.

Exclusion Criteria:

* In addition to exclusion criteria of the parent WARRIOR trial, key exclusion criteria are:
* Non-adherent with IMT. The parent trial is already powered for non-adherence. In our ancillary trial we have built in an exclusion, from final analysis, of an additional 30% who may be nonadherent with IMT or UC.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: This ancillary sub-study will draw 204 patients from the WARRIOR patient group (4422 women), who have undergone a baseline CTA as part of the WARRIOR trial. From this group, 204 patients most compliant with the medication regimen (intensive medical therapy (IMT) with aspirin, statin, angiotensin-converting enzyme inhibitor, and/or angiotensin receptor blocker) vs. usual care (UC) recommended in their treatment groups will undergo a follow-up coronary CTA.
Sampling Method: Non-Probability Sample
Enrollment: 204 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in atherosclerotic plaque burden and noncalcified plaque composition | 3 years
  Change in atherosclerotic plaque burden (%) and noncalcified plaque composition (%) using Autoplaque plaque analysis software
Change in coronary plaque inflammation (measured as CT attenuation of Pericoronary adipose tissue) | 3 years
  Change in pericoronary artery adipose tissue (PCAT) density (CT attenuation of PCAT, in Hounsfield Units) by Autoplaque plaque analysis software
Change in angina score assessed by the Seattle Angina Questionnaire (SAQ) | 3 years
  Change in angina score quantified by the Seattle Angina Questionnaire (SAQ)

CONTACTS AND LOCATIONS:
Overall Officials: Damini Dey, PhD, Principal Investigator — Cedars-Sinai Medical Center; Balaji Tamarappoo, MD, Principal Investigator — Indiana University
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

REFERENCES:
- [Derived] Tamarappoo B, Wolny R, Tomasino GF, Berman D, Handberg E, Pepine CJ, Lo MC, Budoff M, Shaw L, Shufelt C, Wei J, Gulati M, Merz CNB, Dey D. Design and rationale of the WARRIOR ancillary study for coronary CT angiographic analysis. Am Heart J. 2026 Jan 2;294:107340. doi: 10.1016/j.ahj.2026.107340. Online ahead of print. PMID 41485680

DOCUMENTS (1):
  • Informed Consent Form (2022-06-16): https://cdn.clinicaltrials.gov/large-docs/56/NCT05035056/ICF_000.pdf